CLINICAL TRIAL: NCT04585269
Title: Bright IDEAS-Young Adults: Problem-Solving Skills Training to Reduce Distress Among Young Adults With Cancer
Brief Title: Bright IDEAS - Young Adults Problem-Solving Skills Training
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Memorial Sloan Kettering Cancer Center (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Katie Devine, PhD, MPH, Associate Professor Pediatrics, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2019002928; 1R37CA240807-01A1 (NIH); 131911 (Other: CINJ)
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cancer Patients; Young Adult; Supportive Care
Keywords: Young Adults; Cancer; Supportive Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel randomized controlled trial (RCT) of the intervention versus enhanced usual psychosocial care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright IDEAS-YA (Experimental): Intervention consists of six 45-minute one-on-one sessions between a patient and a trainer, who teaches the Bright IDEAS stepwise approach to problem-solving and guides the participant through solving their own problems using the Bright IDEAS approach and worksheets. In addition, participants in this arm will receive a standardized list of resources from the National Comprehensive Cancer Network (NCCN) adolescent and young adult patient guidelines.
  Interventions: Behavioral: Bright IDEAS-YA
- Enhanced Usual Care (No Intervention): Participants in this arm will receive a standardized list of resources from the National Comprehensive Cancer network (NCCN) adolescent and young adult patient guidelines.

INTERVENTIONS:
Behavioral: Bright IDEAS-YA — Bright IDEAS-YA is a manualized problem-solving skills training intervention conducted by a trainer who teaches the participant the Bright IDEAS stepwise approach to problem-solving and guides the participant through solving their own problems using the Bright IDEAS approach.
  Arms: Bright IDEAS-YA

SUMMARY:
The purpose of this project is to evaluate efficacy of Bright IDEAS, an evidence-based problem-solving skills training (PSST) program, as a supportive care intervention for young adult (YA) cancer patients compared with enhanced usual psychosocial care with 344 young adult patients newly diagnosed with cancer.

DETAILED DESCRIPTION:
Bright IDEAS-YA is a personalized approach to increase problem-solving ability by fostering positive appraisal of problems as solvable challenges that can be overcome and enhancing rational problem-solving skills to systematically work through any problem. Bright IDEAS-YA intervention consists of six 45-minute one-on-one sessions with a trainer who teaches the participant the Bright IDEAS stepwise approach to problem-solving and guides the participant through solving their own problems using the Bright IDEAS approach.

Up to 344 young adult patients newly diagnosed with cancer will be recruited to participate in this multi-site randomized controlled trial, where the Bright IDEAS-YA intervention will be compared with enhanced usual psychosocial care. Efficacy will be evaluated by examining changes in psychosocial outcomes from baseline to post-intervention (3 months) and follow-up (6, 12 and 24 months). The extent to which changes in aspects of problem-solving ability mediate the intervention effects will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Current age 18-39
* Within 4 months of first diagnosis of any cancer
* Cancer being treated with chemotherapy and/or radiation therapy and/or hematopoietic stem cell transplant
* No documented or self-reported cognitive delay or impairment that would prevent completion of survey measures
* English-speaking

Exclusion Criteria:

* Medical crisis or not receiving curative therapy per physician/treatment team report
* Treatment involves surgery only

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 344 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Devine, PhD, MPH, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
A final de-identified data set will be made available to researchers with appropriate qualifications for research purposes upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After conclusion of the study
Access Criteria: Investigators with appropriate credentials

REFERENCES:
- [Derived] Bono MH, Reese S, Levonyan-Radloff K, Donovan KA, Sahler OJZ, Barnett ME, Collins M, Devine KA. "There's a lot of unknowns": a thematic analysis of the experiences of young adults with cancer who died during a psychosocial intervention trial. BMC Palliat Care. 2025 Apr 9;24(1):98. doi: 10.1186/s12904-025-01725-2. PMID 40205419
- [Derived] Devine KA, Ohman-Strickland P, Barnett M, Donovan KA, Thompson LMA, Manne SL, Kearney J, Levonyan-Radloff K, Diaz D, Dugad S, Sahler OJZ. Protocol of a Multisite Randomized Controlled Trial of Bright IDEAS-Young Adults: Problem-Solving Skills Training to Reduce Distress among Young Adults with Cancer. Contemp Clin Trials. 2024 Oct;145:107656. doi: 10.1016/j.cct.2024.107656. Epub 2024 Aug 5. PMID 39111386
- [Derived] Kwok G, Reese S, Dugad S, Donovan KA, Tsui J, Sahler OJZ, Levonyan-Radloff K, Barnett ME, Manne S, Ohman-Strickland P, Devine KA. Factors Associated with COVID-19 Vaccine Uptake Among Adolescents and Young Adults Recently Diagnosed with Cancer. J Adolesc Young Adult Oncol. 2024 Apr;13(2):352-357. doi: 10.1089/jayao.2022.0113. Epub 2022 Nov 11. PMID 36367717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: 2/10/2021- 3/12/24 Recruitment modes: in-person (in clinic), and remote (via email and phone).
Period: Baselined and Randomized
Arm/Group | Bright IDEAS-YA | Enhanced Usual Care
Started | 171 | 173
Completed | 171 | 173
Not Completed | 0 | 0
Period: Intervention
Arm/Group | Bright IDEAS-YA | Enhanced Usual Care
Started | 171 | 173
Completed | 123 | 173
Not Completed | 48 | 0
Not completed — Withdrawal by Subject | 9 | 0
Not completed — Unable to schedule | 15 | 0
Not completed — Started but did not finish (<4 sessions) | 24 | 0
Period: FU Time 2 (3 months)
Arm/Group | Bright IDEAS-YA | Enhanced Usual Care
Started | 162 | 173
Completed | 142 | 154
Not Completed | 20 | 19
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 14 | 17
Not completed — Withdrawal by Subject | 4 | 0
Period: FU Time 3 (6 months) Primary outcomes
Arm/Group | Bright IDEAS-YA | Enhanced Usual Care
Started | 156 | 171
Completed | 134 | 146
Not Completed | 22 | 25
Not completed — Death | 4 | 1
Not completed — Lost to Follow-up | 16 | 24
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bright IDEAS-YA | Enhanced Usual Care | Total
Number analyzed (Participants) | 171 | 173 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.00 (6.62) | 30.58 (5.98) | 30.3 (6.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 60 | 68 | 128
  Female | 111 | 104 | 215
  Non-Binary | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 27 | 64
  Not Hispanic or Latino | 134 | 146 | 280
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 23 | 20 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 21 | 17 | 38
  White | 105 | 117 | 222
  More than one race | 6 | 7 | 13
  Unknown or Not Reported | 15 | 11 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 171 | 173 | 344

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptoms of Depression, as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short-Form (v1.0 8a)
Description: Respondents report symptoms on a 5-point rating scale from 1 "never" to 5 "always" in the past 7 days, with higher scores indicating higher levels of negative affect. A total raw summary score is calculated and then translated into a standardized T-score with a mean of 50 and standard deviation of 10, with higher scores indicating higher symptoms. The change in T-score points from baseline to 6 months will be examined, with positive scores indicating increasing symptoms and negative scores indicating decreasing symptoms.
Time Frame: From Baseline to Time 3 (about 6 months from baseline)
Population: Intent-to-treat analyses included all randomized participants (Intervention n = 171; Control n = 173)
Measure: Mean (95% Confidence Interval); unit: T-score points
Arm/Group | Bright IDEAS-YA | Enhanced Usual Care
Number analyzed (Participants) | 171 | 173
T-score points | -2.92 [-4.14 to -1.69] | 0.31 [-0.86 to 1.49]
Statistical Analysis 1: Comparison: Bright IDEAS-YA vs Enhanced Usual Care; Test type: Superiority — Testing for a difference between arms; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.23, 95% CI 2-sided [-4.93 to -1.53]

2. Primary Outcome: Change in Symptoms of Anxiety, as Measured by the PROMIS Anxiety Short-Form (v1.0 8a)
Description: as for outcome 1
Time Frame: From Baseline to Time 3 (about 6 months from baseline)
Population: Intent-to-treat analyses included all randomized participants (Intervention n = 171; Control n = 173)
Measure: Mean (95% Confidence Interval); unit: T-score points
Arm/Group | Bright IDEAS-YA | Enhanced Usual Care
Number analyzed (Participants) | 171 | 173
T-score points | -2.21 [-3.38 to -1.04] | 0.22 [-0.90 to 1.34]
Statistical Analysis 1: Comparison: Bright IDEAS-YA vs Enhanced Usual Care; Test type: Superiority — Testing for a difference between arms; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -2.43, 95% CI 2-sided [-4.05 to -0.81]

3. Primary Outcome: Change in Functional Assessment of Cancer Therapy - General (FACT-G v4)
Description: This 27-item measures health-related quality of life and yields an overall General Total score and four subscales: Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB) and Functional Well-Being (FWB). Respondents rate each item on 5-point Likert scale from 0 (not at all) to 4 (very much) in the past 7 days, where higher numbers indicate higher health state. Each scale is a summary of responses, ranging from 0 to 28 for PWB, SWB, and FWB, 0 to 24 for EWB, and 0 to 108 for General Total.
Time Frame: From Baseline to Time 3 (about 6 months from baseline)
Population: Intent-to-treat analyses included all randomized participants (Intervention n = 171; Control n = 173).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Bright IDEAS-YA | Enhanced Usual Care
Number analyzed (Participants) | 171 | 173
score on a scale | 6.06 [3.85 to 8.27] | 2.66 [0.55 to 4.78]
Statistical Analysis 1: Comparison: Bright IDEAS-YA vs Enhanced Usual Care; Test type: Superiority — Testing for a difference between arms; p = 0.029, Mixed Models Analysis; Mean Difference (Final Values) = 3.40, 95% CI 2-sided [0.34 to 6.45]

4. Secondary Outcome: Symptoms of Depression, as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short-Form (v1.0 8a)
Description: Respondents report symptoms on a 5-point rating scale from 1 "never" to 5 "always" in the past 7 days, with higher scores indicating higher levels of negative affect. A total raw summary score is calculated and then translated into a standardized T-score with a mean of 50 and standard deviation of 10.
Time Frame: Baseline, Time 2 (about 3 months from baseline), Time 4 (about 12 months from baseline), Time 5 (about 24 months from baseline).
Reporting Status: Not Posted

5. Secondary Outcome: Symptoms of Anxiety, as Measured by the PROMIS Anxiety Short-Form (v1.0 8a)
Description: as for outcome 4
Time Frame: as for outcome 4
Reporting Status: Not Posted

6. Secondary Outcome: Functional Assessment of Cancer Therapy - General (FACT-G v4)
Description: as for outcome 3
Time Frame: as for outcome 4
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Comprehensive Score for Financial Toxicity (COST)
Description: Those who indicate financial responsibility will respond to the full 11-item scale of financial toxicity associated with cancer treatment. Respondents rate each item on a 5-point Likert scale from 0 (not at all) to 4 (very much) in the past 7 days. The measure yields a total summary score, with higher scores indicating greater financial strain.
Time Frame: Baseline, Time 4 (about 12 months from baseline), Time 5 (about 24 months from baseline).
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Unmet Needs and Concerns Measured by the Adolescent and Young Adult Oncology Screening Tool (Adapted Version - Young Adults)
Description: Participants first rate their distress on a 0-10 scale. Higher score indicates higher distress. Next, they are asked to check off areas of concern from the past week, including practical (e.g., housing arrangements, work, bills, transportation), family (e.g., parents, siblings, partner), emotional (e.g., sadness, isolation, guilt), social (e.g., isolation from friends, missing important events), physical (e.g., body image, sexual concerns, sleeping difficulty), and informational (e.g., understanding information, feeling involved in decision-making) needs. A total score from 0 to 51 is calculated.
Time Frame: Baseline, Time 2 (about 3 months from baseline), Time 3 (about 6 months from baseline), Time 4 (about 12 months from baseline), Time 5 (about 24 months from baseline).
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S)
Description: This 25-item self-report measure of five theoretically-important constructs of everyday problem-solving, including positive problem orientation, negative problem orientation, rational problem-solving style, impulsive/carelessness style, and avoidant style. Respondents answer each item on 5-point Likert scale from 0 (not at all true of me) to 4 (extremely true of me). Summary scores ranging from 0-20 are computed for each subscale, as well as an overall score. A higher Total score indicates better problem-solving ability.
Time Frame: as for outcome 8
Reporting Status: Not Posted

10. Other Pre Specified Outcome: PROMIS Social Isolation - Short Form 4a
Description: This four-item measure assesses perceptions of social isolation on a 5-point scale from 1 (never) to 5 (always) in the past 7days. Higher scores indicating higher levels of perceived isolation.
Time Frame: as for outcome 8
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Support Services Received
Description: Participants will check whether they have used or received services in the following categories: psychosocial support, informational and practical support, fertility or sexual health, physical/wellness services and integrative medicine services.
Time Frame: as for outcome 8
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Satisfaction With Intervention Derived From the Multi-Dimensional Treatment Satisfaction Measure
Description: Ten-item scale assesses utility of intervention-specific components (e.g., the user manual, worksheets), attitude towards the intervention, trainer competence, and perceived benefit attributable to the intervention. Participants will answer on a 5 point scale, from 1 (strongly disagree) to 5 (strongly agree) with higher scores indicating higher satisfaction. This measure will be administered at post-intervention to intervention arm only.
Time Frame: Time 2 (about 3 months from baseline).
Population: Intervention Arm only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright IDEAS-YA
Number analyzed (Participants) | 171
score on a scale
  Utility: User manual | 4.02 (0.79)
  Utility: Worksheets | 4.00 (0.82)
  Trainer: Warm and supportive | 4.74 (0.63)
  Trainer: Competent | 4.70 (0.63)
  Attitudes: Sessions' length | 4.37 (0.75)
  Attitudes: Number of sessions | 4.12 (0.90)
  I liked the BrightIDEAS program | 4.37 (0.67)
  Perceived benefit: Effectiveness | 4.26 (0.73)
  Perceived benefit: Helpful | 4.08 (0.85)
  Would recommend to other YA | 4.16 (0.96)

ADVERSE EVENTS:
Time Frame: From Baseline and Randomization, through FU Time 3 (6 months). Adverse event data collection is still ongoing and will be updated upon study completion, and additional adverse event data can be added when they become available.
Description: Study team was notified by Epic or medical record (automatically)
Arm/Group | Bright IDEAS-YA | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 6/171 | 3/173
Serious Adverse Events (participants affected / at risk) | 6/171 | 3/173
Other Adverse Events (participants affected / at risk) | 0/171 | 0/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bright IDEAS-YA (N=171) | Enhanced Usual Care (N=173)
Death due to disease progression (General disorders) | 6 (6) | 3 (3) — Participants' death was due to their disease progression, which can be expected when working with patients with cancer. Death was unrelated to the study, which is evaluating a supportive care problem-solving intervention to reduce distress.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT04585269/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT04585269/ICF_000.pdf